CLINICAL TRIAL: NCT01829100
Title: The Function of Avoidance in Depressed Behavior and a Pilot of Transdiagnostic Behavioral Activation Therapy
Brief Title: Transdiagnostic Behavioral Activation Therapy for Youth Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: The Klingenstein Third Generation Foundation (Other)
Responsible Party: Principal Investigator, Brian Chu, Principal Investigator; Associate Professor, Rutgers University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChuDep2009
Record Dates: First submitted 2013-04-04; First posted 2013-04-11 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Depressive Disorder; Anxiety Disorders
Keywords: Adolescent; Transdiagnostic therapy; Behavioral activation; Exposure therapy; Depressive Disorder; Anxiety Disorders
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Behavioral Activation Therapy (Experimental): Group Behavioral Activation Therapy (GBAT)
  Interventions: Behavioral: Group Behavioral Activation Therapy (GBAT)
- waitlist (No Intervention): 15-week waitlist

INTERVENTIONS:
Behavioral: Group Behavioral Activation Therapy (GBAT) — GBAT consists of 15 weekly, hour-long sessions. The first five group sessions teach four core BA principles: (a) psychoeducation of anxiety and depression, (b) functional analysis and identifying the maintaining role of avoidance, (c) problem solving and approach-oriented decision-making, and (d) graded exposures and behavioral activation. The second five group sessions consist of graded exposures or engagement exercises, where group members take turns practicing skills in role plays and in vivo exposures. Each youth receives two individual meetings (30-45 minutes) after the second and fourth group sessions. The first individual meeting promotes engagement and motivation for the group; the second helps develop the youth's individual avoidance/challenge hierarchy.
  Arms: Group Behavioral Activation Therapy

SUMMARY:
Psychological therapies for depression have demonstrated efficacy, but outcomes are still unsatisfactory, especially in cases with high comorbidity. Depression and anxiety co-occur in up to 69-75% of teens and intensify functional impairment and service use. This study will develop treatment materials for a transdiagnostic Group Behavioral Activation Therapy (GBAT) and conduct a pilot waitlist-controlled school-based study with 35 7th and 8th grade boys and girls with co-occurring depression and anxiety. Multi-reporter, multi-domain assessments will be conducted at initial screening, pre- and post-treatment, and 4-month follow-up. BA is a straightforward, but flexible and robust, therapy that has demonstrated strong results in adults. Current formulations of BA highlight the specific role of avoidance in depressotypic behavior. It presumes that anhedonia, isolation, and negative behaviors associated with depression function to avoid imminent distress even as it blocks access to otherwise available positive reinforcement. This study will therefore employ novel electronic diary technology to obtain Ecological Momentary Assessment and evaluate: (a) the function of avoidance in distinguishing youth with depression (n=35) from a non-clinical comparison group (n=18), and (b) the role of avoidance in mediating treatment gains in participants in the GBAT intervention.

DETAILED DESCRIPTION:
Specific Aims and Hypotheses:

This study will develop treatment materials for a transdiagnostic Group Behavioral Activation Therapy (GBAT). It will then conduct a double-gated screening of middle-school students (N=895) to identify youth with subclinical or clinical DSM-IV-TR anxiety or mood disorders. Eligible youth (N=35) will then participate in a randomized clinical trial of GBAT where 21 will be randomly assigned to GBAT and 14 to a 15-week waitlist period. This addresses critical needs to develop first-line early interventions that are evidence-based and can efficiently address commonly co-occurring problems in settings where treatment is needed most.

Aim 1. To develop treatment materials and test GBAT's feasibility (e.g., recruitment and retention rates, therapist adherence) and acceptability to youth participants (client satisfaction, group cohesion, homework completion).

Aim 2. To estimate initial efficacy of GBAT compared to a waitlist (WL) control in a randomized pilot study with 35 youth (21 assigned to two GBAT groups; 14 assigned to WL). It is hypothesized that GBAT will show greater pre- to post-treatment outcomes on primary (clinical diagnosis, symptom severity) and secondary measures (achievement of target goals, reduced avoidance, social and academic adjustment). Youth who receive GBAT will also show linear improvement on outcome measures from pretreatment through four-month follow-up.

A second major goal of the project is to understand the functional role of avoidance in depression. Participating youth will carry Electronic Diaries (EDs; i.e., ipod touch) throughout the active treatment and follow-up phases and complete twice-daily reports of negative events, emotional and behavioral responses, and perceived function of one's responses. A non-clinical comparison group (n=18) will also carry EDs during a two-week period. Such Ecological Momentary Assessment (EMA) data has been used effectively with youth populations to determine the impact of positive and negative coping responses on depressive symptoms.

Aim 3. The research suggests that depressed youth seek out depressogenic activities and respond less to positive events. Based on EMA data, the study hypothesizes that, compared to non-clinical comparisons: (a) depressed youth will identify more events as negative during the day, (b) depressed youth will respond with greater negativity than non-depressed youth, (c) the coping strategies used will be more avoidant or aimed at disengagement, and (d) the function of these strategies will be to minimize distress and conflict. Furthermore, youth who receive GBAT, compared to WL participants, will demonstrate increased ratio of engagement-based to avoidance-based coping strategies from pre- to post-treatment and 4-mo FU.

ELIGIBILITY:
Inclusion Criteria:

* clinical (ADIS CSR ≥ 4) or subclinical (ADIS CSR = 2-3) principal diagnosis of either a DSM-IV-TR unipolar depression disorder (Major Depressive Disorder ([MDD], Minor Depression [MinD], or Dysthymia [Dys]) or
* an anxiety disorder (Generalized Anxiety Disorder [GAD], Social Phobia [SOP], Separation Anxiety [SAD]).

Exclusion Criteria:

* any principal diagnosis other than anxiety or depression or parent report of mental retardation,
* pervasive developmental disorder,
* schizophrenia, or
* bipolar disorder, or
* report of past-year hospitalization for a suicide attempt. Concurrent use of antidepressant or anxiolytic medications was permitted as long as dosage was stable for at least four weeks and the family intended to maintain the dose.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 895 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Diagnosis via the Anxiety Disorders Interview Schedule-IV-TR (ADIS-IV-TR) | Change from baseline (pretreatment) diagnosis at 15 weeks
  ADIS-IV-TR is a semi-structured interview that assesses presence and severity of DSM-IV-TR diagnoses, including parent, child, and consensus diagnosis. Impairment (Clinician's Severity Rating; CSR) is rated per disorder on a 0 (not at all) to 8 (debilitating) scale where 4 represents clinical threshold. The ADIS-IV-TR is administered at pretreatment, posttreatment, and 4-mo FU.

SECONDARY OUTCOMES:
Change in Children's Depression Rating Scale-Revised (CDRS-R) | Change from baseline (pretreatment) symptoms at 31 weeks
  CDRS-R is a clinician-administered interview assessing depression severity over the past week, covering academic, social, health and cognitive functioning, and has been shown to be sensitive to treatment effects. The CDRS-R is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Children's Depression Rating Scale-Revised (CDRS-R) | Change from baseline (pretreatment) symptoms at 15 weeks
  CDRS-R is a clinician-administered interview assessing depression severity over the past week, covering academic, social, health and cognitive functioning, and has been shown to be sensitive to treatment effects. The CDRS-R is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Diagnosis via the Anxiety Disorders Interview Schedule-IV-TR (ADIS-IV-TR) | Change from baseline (pretreatment) diagnosis at 31 weeks
  ADIS-IV-TR is a semi-structured interview that assesses presence and severity of DSM-IV-TR diagnoses, including parent, child, and consensus diagnosis. Impairment (Clinician's Severity Rating; CSR) is rated per disorder on a 0 (not at all) to 8 (debilitating) scale where 4 represents clinical threshold. The ADIS-IV-TR is administered at pretreatment, posttreatment, and 4-mo FU.

OTHER OUTCOMES:
Change in Clinical Global Impression - Severity (CGI-S) | Change from baseline (pretreatment) impairment at 31 weeks
  CGI-S is a widely-used clinician rating scale of symptom severity from 0 (no illness) to 6 (extremely severe) and is sensitive to treatment effects. The CGI-S is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Screen for Child Anxiety Related Emotional Disorders (SCARED). | Change from baseline (pretreatment) symptoms at 31 weeks.
  SCARED is a 41-item self-report scale of anxiety symptoms experienced in the past three months. Total scores above 25 are indicative of an anxiety disorder. Previous research indicates strong discriminant and convergent validity. The SCARED is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Center for Epidemiologic Studies-Depression Scale (CES-D). | Change from baseline (pretreatment) symptoms at 31 weeks
  CES-D is a 20 item self-report scale of depressive symptoms experienced over the past week. Total scores ≥ 21 predict significant presence of depression over the next year. Good psychometric data exist for use of the CES-D with adolescents. The CES-D is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Strengths and Difficulties Questionnaire (SDQ) | Change from baseline (pretreatment) impairment at 31 weeks.
  SDQ is a 25-item behavioral screening questionnaire assessing five emotional and behavioral domains and has good psychometric properties (e.g., reliability and convergent validity). SDQ is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Behavioral Activation of Depression Scale - Adolescent (BADS-A) | Change from baseline (pretreatment) activation at 31 weeks
  BADS-A is a 26-item adaptation of the adult BADS and assesses behavioral activation and avoidance. BADS-A was adapted for the current study to reflect developmentally appropriate reading level and concepts. The BADS and BADS-A have strong psychometric properties including reliability and predictive validity. BADS-A is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Child Automatic Thoughts Scale (CATS) | Change from baseline (pretreatment) negative thinking at 31 weeks
  CATS is a 40-item child-report measure designed to assess negative self-statements, and has demonstrated good reliability and discriminant validity. The CATS is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Clinical Global Impression - Severity (CGI-S) | Change from baseline (pretreatment) impairment at 15 weeks
  CGI-S is a widely-used clinician rating scale of symptom severity from 0 (no illness) to 6 (extremely severe) and is sensitive to treatment effects. The CGI-S is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Screen for Child Anxiety Related Emotional Disorders (SCARED). | Change from baseline (pretreatment) symptoms at 15 weeks.
  SCARED is a 41-item self-report scale of anxiety symptoms experienced in the past three months. Total scores above 25 are indicative of an anxiety disorder. Previous research indicates strong discriminant and convergent validity. The SCARED is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Center for Epidemiologic Studies-Depression Scale (CES-D). | Change from baseline (pretreatment) symptoms at 15 weeks
  CES-D is a 20 item self-report scale of depressive symptoms experienced over the past week. Total scores ≥ 21 predict significant presence of depression over the next year. Good psychometric data exist for use of the CES-D with adolescents. The CES-D is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Strengths and Difficulties Questionnaire (SDQ) | Change from baseline (pretreatment) impairment at 15 weeks.
  SDQ is a 25-item behavioral screening questionnaire assessing five emotional and behavioral domains and has good psychometric properties (e.g., reliability and convergent validity). SDQ is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Behavioral Activation of Depression Scale - Adolescent (BADS-A) | Change from baseline (pretreatment) activation at 15 weeks
  BADS-A is a 26-item adaptation of the adult BADS and assesses behavioral activation and avoidance. BADS-A was adapted for the current study to reflect developmentally appropriate reading level and concepts. The BADS and BADS-A have strong psychometric properties including reliability and predictive validity. BADS-A is administered at pretreatment, posttreatment, and 4-mo FU.
Change in Child Automatic Thoughts Scale (CATS) | Change from baseline (pretreatment) negative thinking at 15 weeks
  CATS is a 40-item child-report measure designed to assess negative self-statements, and has demonstrated good reliability and discriminant validity. The CATS is administered at pretreatment, posttreatment, and 4-mo FU.

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Chu, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States